CLINICAL TRIAL: NCT00584766
Title: Intensive Combination Chemotherapy With Autologous Bone Marrow Rescue for Metastatic Breast Cancer After Intitial Cytoreduction With Standard Agents: A Phase II Study
Brief Title: Intensive Combo Chemo With Autologous BM Rescue for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: George Selby, University of Oklahoma Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU 8701; OU 8701
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: High-dose chemotherapy

INTERVENTIONS:
Procedure: High-dose chemotherapy — Cyclophosphamide 500 mg/m2 IV day 1; Doxorubicin 30 mg/m2 IV Day 1; Methotrexate 300 mg/m2 IV Day 8;5-FU 500 mg/m2 IV day 8; leucovorin 20 mg po q 6 h x 6 doses, day 9- cycles repeated q 21 days

SUMMARY:
To determine the therapeutic efficacy of high-dose cyclophosphamide and BCNU with autologous bone marrow transplantation after initial tumor cytoreduction for patients with receptor-negative metastatic breast carcinoma and to determine the optimal timing of CyBCNU-ABMT after initial development of metastatic breast carcinoma

ELIGIBILITY:
Inclusion Criteria:

* breast carcinoma at first clinical evidence of metastatic disease
* must have measurable disease by physical exam, x-ray, or scan
* Age < or equal to 55
* performance status 0-2

Exclusion Criteria:

* can't have had more than one prior chemotherapy regimen
* can't have had concurrent hormonal therapy
* no brain metastases
* no previous pelvic radiation
* no history of another malignancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 1987-10; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Quality of maximal response; time to initial disease progression; and overall survival | undetermined

SECONDARY OUTCOMES:
to determine the optimal timing of CyBCNU-ABMT after initial development of metastatic breast cancer | undetermined

CONTACTS AND LOCATIONS:
Overall Officials: George Selby, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States